CLINICAL TRIAL: NCT00869011
Title: Effects of Physical Activity on the Endothelial and Cardiac Function of Patients With Renal Cell Carcinoma Receiving a Thyrosine Kinase Inhibitor (Sunitinib)
Brief Title: Exercise for Patients With Renal Cell Cancer Receiving Sunitinib
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Pfizer (Industry)
Responsible Party: PD Dr. Fernando C. Dimeo, Dept. of Sports Medicine, Charité Universitätsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SUIR8687
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Cancer; renal cell carcinoma; fatigue; exercise
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Fatigue; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Exercise
  Interventions: Other: Endurance exercise
- 2 (No Intervention): No structured exercise program

INTERVENTIONS:
Other: Endurance exercise — Endurance exercise, 3 times weekly for 35-45 minutes, 12 weeks.
  Arms: 1

SUMMARY:
In this randomized, controlled trial the investigators evaluate the effects of an exercise program lasting for 12 weeks on the physical performance, the cardiovascular function (24h blood pressure, rest blood pressure and hear function) and the fatigue and mood of patients with renal cell carcinoma undergoing a therapy with Sunitinib.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years
* Understanding of written German
* Treatment with Sunitinib
* Ability to walk

Exclusion Criteria:

* Cardiovascular, pulmonary or osteoarticular disease which can be aggravated by exercise
* BMI < 18 or > 30

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 12 weeks

SECONDARY OUTCOMES:
VO2max | 12 weeks
Systolic and diastolic blood pressure (24 h) | 12 weeks
Depression score | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Section Sports Medicine, Charité Universitätsmedizin Berlin, Hindenburgdamm 30, Berlin, State of Berlin, Germany